CLINICAL TRIAL: NCT06236698
Title: Accuracy of 24-hour Urinary Aldosterone Testing in Diagnosing Primary Aldosteronism and Analysis of Drug Interference Factors
Brief Title: The Diagnostic Performance of 24-hour Urinary Aldosterone for Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: Zhiming Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhiming Zhu, Professor, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: The value of 24h UA
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Primary Aldosteronism; Hypertension
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Essential hypertension: Adult patients meet the 2018 Chinese guidelines for prevention and treatment of hypertension for a diagnosis of essential hypertension but without other obvious features of PA.
  Interventions: Diagnostic Test: 24-hour urinary aldosterone measurement
- Primary aldosteronism: Adult patients meet the Endocrine Society Clinical Practice Guidelines for a diagnosis of primary aldosteronism.
  Interventions: Diagnostic Test: 24-hour urinary aldosterone measurement

INTERVENTIONS:
Diagnostic Test: 24-hour urinary aldosterone measurement — Collect 24-hour urine sample from each participant and complete the detection of urinary aldosterone content.

SUMMARY:
This is an observational study to define the cut-off value of 24-hour urinary aldosterone for diagnosing primary aldosteronism in hypertensive patients in our center. Plasma aldosterone and renin measurements are subject to significant intra-individual variability, including variation related to posture, time of day and sodium balance. Aldosterone secretion is not constant and may be subject to diurnal variation. As such one-off testing of ARR, does not consider the salt status of the individual necessitating repetition of tests to ensure false negative or false positive test results are ruled out. The value of accumulated aldosterone in a 24-hour sample has the advantage that it does not depend on circadian variation. This study will help establish the positivity rates of 24-hour urine aldosterone, and test the robustness of current standard guidelines for primary aldosteronism screening and case confirmation.

Previous studies reported that primary aldosteronism is associated with a higher risk of CV complications and a higher prevalence of target organ damage. Also, previous studies reported on the association of echocardiographic parameters with circulating or urinary aldosterone. Therefore, we intent to investigate the independent associations of different target organ damage with the urinary excretion of aldosterone.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and above.
2. Meets the 2018 Chinese guidelines for prevention and treatment of hypertension for a diagnosis of hypertension with an age of onset of hypertension between 18-80 years.
3. Meets the Endocrine Society Clinical Practice Guidelines for a diagnosis of primary aldosteronism with an age of onset of hypertension between 18-80 years.

Exclusion Criteria:

1. Other causes of secondary hypertension, including renal hypertension, renovascular hypertension and adrenal hypertension (i.e., pheochromocytoma and Cushing syndrome).
2. Urine output less than 400ml per day.
3. Severe renal insufficiency with a glomerular filtration rate < 60 mL/min/1.73 m2.
4. lack of 24-h urinary aldosterone data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We recruited hypertensive individuals who were hospitalized in the Department of Hypertension and Endocrinology of Daping Hospital from April 2022 to October 2024.
  Group 1: Adult patients meet the 2018 Chinese guidelines for prevention and treatment of hypertension for a diagnosis of essential hypertension but without other obvious features of primary aldosteronism.
  Group 2: Adult patients meet the Endocrine Society Clinical Practice Guidelines for a diagnosis of primary aldosteronism.
Sampling Method: Non-Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
The cut-off value of 24-hour urinary aldosterone for distinguishing primary aldosteronism from primary hypertension. | 2 years
  This study will define the cut-off value of 24-hour urinary aldosterone for identifying patients with primary aldosteronism in hypertensive patients.

SECONDARY OUTCOMES:
Impacts of antihypertensive medications on 24-h urinary aldosterone levels | 2 years
  Antihypertensive drugs are usually stopped prior to diagnostic testing since they affect the physiological renin-angiotensin-aldosterone system. It is frequently unsafe and impractical to stop taking all conflicting antihypertensive drugs, especially in patients with severe hypertension. The impact of antihypertensive drugs on 24-hour urinary aldosterone, however, has not yet been documented. We tried to investigate how antihypertensive drugs affected 24-hour urine aldosterone levels in this investigation.
The relationship between 24-hour urinary aldosterone and target organ damage in hypertension. | 2 years
  This study will gain futher insight in the association between different target organ damage and the urinary excretion of aldosterone. We will try to find out the reationship between urinary aldosterone and renal function indicators, including eGFR and Urinary microalbumin, and cardiac function indicators, including IVST and PWT.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Zhu, MD, Study Chair — Department of Hypertension and Endocrinology, Daping Hospital, Army Medical University
Locations (1):
- China Chongqing The third hospital affiliated to the Third Millitary Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided